CLINICAL TRIAL: NCT03594682
Title: Optimizing the Therapeutic Dose of Apatinib Mesylate Tablets in Patients With Lung Cancer by Dose Titration：A Real World Exploratory Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beijing Chest Hospital (Other)
Responsible Party: Principal Investigator, Ying Hu, Vice Director,Department of oncology, Beijing Chest Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HB-B001
Record Dates: First submitted 2018-06-24; First posted 2018-07-20 (Actual); Last update posted 2018-07-20 (Actual); Status verified 2018-06

CONDITIONS: NSCLC Stage IV; NSCLC Stage IIIB
Keywords: Apatinib,NSCLC,Dose titration
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Methods; Therapeutics

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- dose titration group (Experimental): First of all, according to the patient's weight and ECOG score, patients were divided into three groups（the initial dose of 250 mg qd,250 mg/500 mg qd by turns, 500 mg qd）. in two weeks, if the patient who is intolerant of the initial dose,250mg qod,250mg qd ,250mg qd was selected. if the patient can tolerate the dose well,a high-dose was given,and the maximum dose does not exceeding 750mg qd.
  Interventions: Other: Intervention/treatment
- non-titration group (Active Comparator): Patients were given 750mg qd apatinib until disease progression or intolerance
  Interventions: Other: Intervention/treatment

INTERVENTIONS:
Other: Intervention/treatment — experimentalgroup initial dose：
  1. 250mg qod
  2. 250mg qd/500mg qd by turn
  3. 500mg qd control group： 750mg qd

SUMMARY:
The purpose of the study is to evaluate the safety and efficacy of two different administration methods of apatinib in NSCLC patients.

DETAILED DESCRIPTION:
1. Aged ≥18；
2. Locally advanced/metastatic non-small lung cancer (IIIb/IV) confirmed by pathology with measurable lesions；
3. Patients with wild type EGFR/ALK must received two kinds of systemic chemotherapy before；Patients with EGFR mutation positive had experienced treatment failure with TKI in first line and Chemotherapy in second line ；
4. ECOG：0-4；
5. The subjects were treated with other drugs has been restored (NCI CTCAE version 4.0 class 1 or less), which accept nitroso urea or mitomycin interval 6 weeks or more; Accept other cytotoxic drugs, bevacizumab (Avastin) (except local palliative radiotherapy), radiotherapy or surgery four weeks or more. EGFR TKI ≥2 weeks; Main organs function is normal；
6. Fertile woman must perform a pregnancy test (serum or urine) 7 days before screened, or voluntarily adopt proper methods of contraception during the observation period and 8 week after the last given apatinib. For man, surgical sterilization should be performed, or voluntarily adopt proper methods of contraception during the observation period and 8 week after the last given apatinib；
7. Patients voluntarily entered the study and signed informed consent form (ICF).

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥18；
2. Locally advanced/metastatic non-small lung cancer (IIIb / IV) confirmed by pathology with measurable lesions ；
3. Patients with wild type EGFR/ALK must received two kinds of systemic chemotherapy before；Patients with EGFR mutation positive had experienced treatment failure with TKI in first line and Chemotherapy in second line ；
4. ECOG：0-4；
5. The subjects were treated with other drugs has been restored (NCI CTCAE version 4.0 class 1 or less), which accept nitroso urea or mitomycin interval 6 weeks or more; Accept other cytotoxic drugs, bevacizumab (Avastin) (except local palliative radiotherapy), radiotherapy or surgery four weeks or more. EGFR TKI ≥2 weeks; Main organs function is normal；
6. Fertile woman must perform a pregnancy test (serum or urine) 7 days before screened, or voluntarily adopt proper methods of contraception during the observation period and 8 week after the last given apatinib. For man, surgical sterilization should be performed, or voluntarily adopt proper methods of contraception during the observation period and 8 week after the last given apatinib；
7. Patients voluntarily entered the study and signed informed consent form (ICF).

Exclusion Criteria:

1. brain MRI, CT or venography confirmed that there are brain hemorrhage symptoms；
2. Tumor invade big vessels or close to big vessels (less than 5mm)；
3. Patients with uncontrollable hypertension (systolic blood pressure> 140 mmHg, diastolic blood pressure> 90 mmHg, despite optimal drug therapy).；
4. Patients with with grade Ⅱ myocardial ischemia or myocardial infarction, poor control of arrhythmias (including QTc interval male ≥ 450 ms, female ≥470 ms)；
5. Abnormal coagulation (INR>1.5 or PT>ULN+4, or APTT>1.5 ULN), bleeding tendency or receiving coagulation therapy
6. Urine protein≥++, or urine protein in 24 hours≥1.0g
7. CTCAE 2 degrees or more peripheral neuropathy, except the trauma;
8. Unhealed bone fracture or wound for long time；
9. Patients who received systemic antibiotic treatment of serious infections;
10. Decompensated diabetes or high dose of glucocorticoid treatment other banned disease;
11. Patients with active hepatitis B virus or hepatitis c virus infection；
12. Patients with obvious factors affecting absorption of oral drugs, such as difficulties in swallowing, chronic diarrhea and intestinal obstruction, etc.
13. Received big surgery, had bone fracture or ulcer in 4 weeks.
14. Within 6 weeks before random severe weight loss (> 10%);
15. Patients who experienced bleeding symptoms of clinical significance within 3 months before screening, or with confirmed bleeding tendency such as hemorrhage of digestive tract, hemorrhagic gastric ulcer, baseline occult blood in stool ++ and above, or vasculitis, etc；
16. Random 12 months before the artery/vein thrombosis events, such as cerebrovascular accident (including transient ischemic attack, cerebral hemorrhage, cerebral infarction), deep vein thrombosis and pulmonary embolism, etc.；
17. Known history of hypersensitivity to apatinib or any of it components.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Estimated)
Dates: Start 2018-08 (Estimated); Primary Completion 2019-07 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
duration of treatment | two years
  time from take apatinib to withdrawal from experiment due to adverse reaction of apatinib

CONTACTS AND LOCATIONS:
Overall Officials: Li Baolan, Study Director — Beijing Chest Hospital